CLINICAL TRIAL: NCT03192137
Title: A Phase 3, Randomized, Multicenter, Double-masked Study to Compare the Ocular Safety, Tolerability, and Efficacy of ISV-305 (0.1% Dexamethasone in DuraSite® 2) to DuraSite 2 Vehicle for the Treatment of Inflammation and Pain Associated With Cataract Surgery
Brief Title: Study to Evaluate ISV-305 Compared to Vehicle for Treatment of Inflammation and Pain Associated With Cataract Surgery
Acronym: ISV-305
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-13-305-002
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Results first posted 2020-06-29 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Inflammation and Pain Associated With Cataract Surgery
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ISV-305 (Experimental): 0.1% dexamethasone in DuraSite® 2
  Interventions: Drug: ISV-305
- Vehicle (Placebo Comparator): DuraSite® 2 Vehicle
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: ISV-305 — Dexamethasone in DuraSite® 2 twice daily for 16 days
  Arms: ISV-305
Other: Vehicle — Vehicle twice daily for 16 days
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the ocular safety, tolerability, and efficacy of ISV-305 (dexamethasone in DuraSite® 2) compared with Vehicle in the treatment of inflammation and pain associated with cataract surgery.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the ocular safety, tolerability, and efficacy of topical administration of ISV-305 (0.1% dexamethasone in DuraSite® 2) compared with Vehicle when dosed twice daily for 1 day prior to surgery, the day of surgery and 14 days post cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 17 years of age
* Are scheduled for uncomplicated unilateral cataract surgery
* Signature of the subject or parent(s) or legally authorized representative on the Informed Consent Form, and when appropriate the minor's assent in accordance with local regulations
* Are willing and able to follow all instructions and attend all study visits
* Are willing to avoid disallowed medication for the duration of the study
* If female is of childbearing potential, agree to and submit a urine sample for pregnancy testing (prior to enrollment and at the end of the study) and use effective contraception for the duration of the study
* Male subjects whose female partners are not post-menopausal must agree to one of the following: 1) completely abstain from sexual intercourse, 2) use a barrier method (condoms) with spermicide during sexual intercourse for the duration of the study, 3) provide documentation for having had a vasectomy (with documented infertility)
* Additional inclusion criteria also apply

Exclusion Criteria:

* Have known sensitivity or poor tolerance to any component of the study drugs
* Have any sign of iritis or scleritis in the study eye
* Have an acute ocular infection (bacterial, viral or fungal) or active ocular inflammation in the study eye
* Have any active or chronic/recurrent ocular or systemic disease that is uncontrolled and likely to affect wound healing (e.g., diabetes mellitus, systemic connective tissue disease, severe atopic disease)
* Have known blood dyscrasia or bone marrow suppression
* Have any active corneal pathology in the study eye
* Have had radial keratotomy, corneal transplant, or LASIK in the study eye within the last 2 years
* Be currently pregnant, nursing, or planning a pregnancy; or have a positive urine pregnancy test
* Have prior (within 30 days of beginning study treatment) or anticipated concurrent use of an investigational drug or device
* Have a condition or a situation which, in the investigator's opinion, may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation
* Use of any medication the investigator feels may interfere with the study parameters
* Additional exclusion criteria also apply

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ISV-305: ISV-305 was administered as a topical ophthalmic formulation of 0.1% dexamethasone in DuraSite® 2 vehicle (InSite Vision's drug delivery system) twice daily (one drop in the morning and one drop in the evening) for 16 days.
- Vehicle: Vehicle (DuraSite® 2 vehicle) was administered as a matching topical ophthalmic formulation without dexamethasone twice daily (one drop in the morning and one drop in the evening) for 16 days.
Period: Overall Study
Arm/Group | ISV-305 | Vehicle
Started | 173 | 87
Completed | 123 | 29
Not Completed | 50 | 58
Not completed — Adverse Event | 10 | 11
Not completed — Physician Decision | 1 | 0
Not completed — Lack of Efficacy | 20 | 37
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Protocol Violation | 4 | 3
Not completed — Surgery Cancelled | 4 | 1
Not completed — Other - Various Administrative Reasons | 8 | 3

BASELINE CHARACTERISTICS:
Population: Demographics were summarized for the Safety Population which included all randomized participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | ISV-305 | Vehicle | Total
Number analyzed (Participants) | 158 | 80 | 238
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (7.15) | 68.5 (9.37) | 68.2 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 43 | 137
  Male | 64 | 37 | 101
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 5 | 15
  White | 141 | 72 | 213
  Mixed | 0 | 1 | 1
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Anterior Chamber Cell (ACC) Grade 0 in Study Eye at Day 15 (Last Observation Carried Forward) in the Modified Intent to Treat (mITT) Population
Description: Biomicroscopic measurement of anterior chamber cells was conducted in the surgery eye (study eye) by the same examiner from visit to visit whenever possible. A slit-lamp biomicroscope was used at x16 magnification with a 1 x 1 mm oblique high-intensity beam. Two cell counts were summed and divided by 2 to determine an average final anterior chamber cell count. This final cell count was converted to a grade: Grades 0, 1, 2, 3, 4 were assigned for cell counts of 0, 1 to 10, 11 to 20, 21 to 50, and > 50, respectively. If the averaged count fell between two grades, the higher grade was selected (e.g., if the two counts were 10 and 11, the average of 10.5 fell into Grade 2). Missing anterior chamber cell grade at Day 15 was imputed by last non-missing scheduled post-baseline anterior chamber cell grade assessed prior to Day 15 (last observation carried forward).
Time Frame: Day 15
Population: mITT Population - included randomized participants who underwent cataract surgery, received at least one dose of ISV-305 or vehicle, and had at least one post-surgery efficacy assessment (ACC or VAS). Participants who received rescue medications were included in the mITT Population, but were treated as failures.
Measure: Number; unit: participants
Arm/Group | ISV-305 | Vehicle
Number analyzed (Participants) | 144 | 72
participants
  0 (did not receive rescue therapy) | 69 | 16
  0 (received rescue therapy) | 0 | 0
  1 | 64 | 30
  2 | 5 | 10
  3 | 6 | 12
  4 | 0 | 4
Statistical Analysis 1: Comparison: ISV-305 vs Vehicle; Test type: Superiority — Statistical hypotheses testing for the primary efficacy endpoint was two-sided and performed using a significance (alpha) level of 0.05; p = 0.0005, Chi-squared, Corrected — P-values were from a Chi-Square test (with continuity correction) of differences between treatments in the proportion of participants with anterior chamber cells Grade 0 who did not receive rescue medication versus all other grades combined; A Fisher's exact test was used if 1 or more of the cells had an expected frequency of ≤ 5

2. Secondary Outcome: Proportion of Participants Who Achieved a Pain Score of 0 on the Visual Analog Scale (VAS) for Each Post-surgical Assessment
Description: Eye pain/discomfort in the study eye was evaluated at every visit except Visit 2 (Surgery; Day 0) using a VAS, scoring from 0 to 100 using a mark on a 100 mm line (0 = absent; 100 = maximum). Participants were asked to rate the feeling of the symptom in the study eye from absent to extreme by moving a slide on the side of the scale to align with images of descriptive faces.
Time Frame: Day 1 to Day 29
Population: mITT Population - included randomized participants who underwent cataract surgery, received at least one dose of ISV-305 or vehicle, and had at least one post-surgery efficacy assessment (ACC or VAS). Participants who received rescue medications were included in the mITT Population but were treated as failures.
Measure: Number; unit: Participants
Arm/Group | ISV-305 | Vehicle
Number analyzed (Participants) | 156 | 77
Participants
  Pain Score of 0 on Day 1 | 103 | 29
  Pain Score of 0 on Day 8 | 133 | 44
  Pain Score of 0 on Day 15 | 137 | 49
  Pain Score of 0 on Day 18 | 129 | 50
  Pain Score of 0 on Day 29 | 135 | 51
Statistical Analysis 1: Comparison: ISV-305 vs Vehicle; Statistical analysis of proportion of participants who achieved a pain score of 0 on the VAS on Day 1; Test type: Superiority — Statistical hypotheses testing for the secondary efficacy endpoints were two-sided and performed using a significance (alpha) level of 0.05; p < 0.0001, Chi-squared, Corrected — P-values were from a Chi-Square test (with continuity correction); A Fisher's exact test was used if 1 or more of the cells had an expected frequency of ≤ 5; Odds Ratio (OR) = 3.217, 95% CI 2-sided [1.823 to 5.675]
Statistical Analysis 2: Comparison: ISV-305 vs Vehicle; Statistical analysis of proportion of participants who achieved a pain score of 0 on the VAS on Day 8; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Chi-squared, Corrected — P-values were from a Chi-Square test (with continuity correction); A Fisher's exact test was used if 1 or more of the cells had an expected frequency of ≤ 5; Odds Ratio (OR) = 4.337, 95% CI 2-sided [2.305 to 8.161]
Statistical Analysis 3: Comparison: ISV-305 vs Vehicle; Statistical analysis of proportion of participants who achieved a pain score of 0 on the VAS on Day 15; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Chi-squared, Corrected — P-values were from a Chi-Square test (with continuity correction); A Fisher's exact test was used if 1 or more of the cells had an expected frequency of ≤ 5; Odds Ratio (OR) = 4.120, 95% CI 2-sided [2.113 to 8.033]
Statistical Analysis 4: Comparison: ISV-305 vs Vehicle; Statistical analysis of proportion of participants who achieved a pain score of 0 on the VAS on Day 18; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0043, Chi-squared, Corrected — P-values were from a Chi-Square test (with continuity correction); A Fisher's exact test was used if 1 or more of the cells had an expected frequency of ≤ 5; Odds Ratio (OR) = 2.580, 95% CI 2-sided [1.380 to 4.822]
Statistical Analysis 5: Comparison: ISV-305 vs Vehicle; Statistical analysis of proportion of participants who achieved a pain score of 0 on the VAS on Day 29; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0005, Chi-squared, Corrected — P-values were from a Chi-Square test (with continuity correction); A Fisher's exact test was used if 1 or more of the cells had an expected frequency of ≤ 5; Odds Ratio (OR) = 3.277, 95% CI 2-sided [1.695 to 6.335]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from the date of signing the consent form to the date of completion of the participant's final visit (Day 29). Ongoing AEs were followed beyond the final study visit at the discretion of the investigator.
Description: Treatment-emergent adverse events were summarized for the Safety Population, which included all randomized participants who received at least one dose of study treatment (i.e., 158 and 80 subjects in the ISV-305 and Vehicle arms, respectively).
Arm/Group | ISV-305 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/158 | 0/80
Serious Adverse Events (participants affected / at risk) | 3/158 | 0/80
Other Adverse Events (participants affected / at risk) | 31/158 | 21/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ISV-305 (N=158) | Vehicle (N=80)
Chest pain (General disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ISV-305 (N=158) | Vehicle (N=80)
Iritis (Eye disorders) | 6 | 5
Visual acuity reduced (Eye disorders) | 7 | 2
Eye pain (Eye disorders) | 3 | 4
Cystoid macular oedema (Eye disorders) | 2 | 3
Eye inflammation (Eye disorders) | 1 | 4
Foreign body sensation in eyes (Eye disorders) | 2 | 3
Visual impairment (Eye disorders) | 4 | 1
Intraocular pressure increased (Investigations) | 10 | 2
Headache (Nervous system disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit the manuscript of any journal article, abstract or other presentation arising from an InSite Vision-sponsored clinical investigation to InSite Vision for editorial review prior to submission for publication or presentation. At the sponsor's request, if proprietary information is to be disclosed, proposed publications or presentations will be delayed until appropriate patent applications and/or legal documents of a similar nature have been filed.

DOCUMENTS (2):
  • Study Protocol (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT03192137/Prot_001.pdf
  • Statistical Analysis Plan (2017-12-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT03192137/SAP_002.pdf